CLINICAL TRIAL: NCT01383915
Title: Characterizing the Clinical Risk State for Bipolar Disorder in Adolescents
Brief Title: Clinical Risk State for Bipolar Disorder in Adolescents
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Christoph U. Correll, MD, Principal Investigator, Northwell Health
Other Study IDs: 06-123
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Bipolar Disorder; Schizophrenia
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- inpatients: Youth with a clinical diagnosis of a mood disorder or psychosis spectrum disorder

SUMMARY:
Aim: The purpose of the study is to characterize the at-risk phases preceding a first episode of bipolar disorder and of schizophrenia, and to identify clinical and biological predictors of the disease development.

Hypothesis a: Over 6-24 months, 25% of at-risk youth will develop the full manifestations of Bipolar Disorder (BPD) or schizophrenia.

Hypothesis b: The symptoms utilized for characterizing the at-risk phase of BPD will differentiate between individuals developing BPD and schizophrenia.

DETAILED DESCRIPTION:
Prospective, naturalistic, cohort study aiming to characterizing the bipolar and psychotic prodrome thoroughly with a variety of clinical and biological measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 12-18 years;
2. Sex: male or female;
3. Race/ethnicity: no restrictions;
4. Definite or suspected chart diagnosis of BP-II, BP-NOS, cyclothymia, MDD, depressive disorder NOS, dysthymia or mood disorder NOS, schizophrenifiorm disorder or psychotic disorder NOS;
5. Subject and parent (if subject<18) willing and able to provide written, informed consent/assent.

Exclusion Criteria:

1. Estimated Premorbid IQ < 70;
2. Meets DSM-IV criteria for BP-I or schizophrenia, pervasive developmental disorder, autism spectrum disorders, current substance dependence;
3. History of medical condition known to affect the brain;
4. current group home affiliation.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Inpatients consecutively admitted to the adolescent inpatient unit of the Zucker Hillside Hospital, NY
Sampling Method: Non-Probability Sample
Enrollment: 402 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with development of a bipolar or schizophrenia disorder | within 60 months
  Diagnostic conversion

SECONDARY OUTCOMES:
Psychopathology | within 60 months
  Psychopathology

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Correll, MD, Principal Investigator — The Zucker Hillside Hospital, Feinstein Institute for Medical Research
Locations (1):
- The Zucker Hillside Hospital, NSLIJ, Glen Oaks, New York, United States

REFERENCES:
- [Derived] Gerstenberg M, Hauser M, Al-Jadiri A, Sheridan EM, Kishimoto T, Borenstein Y, Vernal DL, David L, Saito E, Landers SE, Carella M, Singh S, Carbon M, Jimenez-Fernandez S, Birnbaum ML, Auther A, Carrion RE, Cornblatt BA, Kane JM, Walitza S, Correll CU. Frequency and correlates of DSM-5 attenuated psychosis syndrome in a sample of adolescent inpatients with nonpsychotic psychiatric disorders. J Clin Psychiatry. 2015 Nov;76(11):e1449-58. doi: 10.4088/JCP.14m09435. PMID 26646040